CLINICAL TRIAL: NCT03199651
Title: Beating Lung Cancer in Ohio (BLCIO) Protocol
Brief Title: Beating Lung Cancer in Ohio Protocol in Improving Survival in Patients with Stage IV Non-Small Cell Lung Cancer
Acronym: BLCIO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Peter Shields, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: OSU-17070; NCI-2017-00723 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2017-05-26; First posted 2017-06-27 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Cigarette Smoker; Current Smoker; Lung Adenocarcinoma; Squamous Cell Lung Carcinoma; Stage IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung | interventions — Practice Guidelines as Topic; Standard of Care; Smoking Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (UC) (Active Comparator): Patients receive usual care and undergo collection of tumor tissue and blood sample for the repository. Patients who smoke or have recently quit smoking and their household members who smoke may also undergo smoking cessation via usual care or NCCN driven-CTC/DS.
  Interventions: Other: Best Practice; Procedure: Biospecimen Collection; Other: Laboratory Biomarker Analysis; Other: Medical Chart Review; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Behavioral: Smoking Cessation Intervention
- Arm II (AGIT/DS) (Experimental): Patients undergo collection of tumor tissue for analysis using FoundationOne assay and blood sample for analysis using FoundationACT blood circulating tumor DNA assay. Patients who smoke or have recently quit smoking and their household members who smoke may also undergo smoking cessation via usual care or NCCN driven-CTC/DS.
  Interventions: Procedure: Biospecimen Collection; Other: Laboratory Biomarker Analysis; Other: Medical Chart Review; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Behavioral: Smoking Cessation Intervention

INTERVENTIONS:
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
  Arms: Arm I (UC)
Procedure: Biospecimen Collection — Undergo collection of tumor tissue and blood sample for repository
  Arms: Arm I (UC)
Procedure: Biospecimen Collection — Undergo tumor tissue and blood sample for AGIT/DS
  Arms: Arm II (AGIT/DS)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Medical Chart Review — Undergo medical record abstraction
  Other Names: Chart Review
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Behavioral: Smoking Cessation Intervention — Undergo usual care or NCCN-driven CTC/DS
  Other Names: Smoking and Tobacco Use Cessation Interventions

SUMMARY:
This randomized clinical trial studies the Beating Lung Cancer in Ohio protocol in improving survival in patients with stage IV non-small cell lung cancer. The Beating Lung Cancer in Ohio protocol may help in evaluating immunotherapies and targeted therapies that prolong survival, have more favorable toxicity profiles than conventional chemotherapy and impact quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

1a. Establish a 3 month observation period for newly diagnosed stage IV non-small cell lung cancer patients (NSCLC)(n=300), using the statewide research network, documenting usual care (UC) practices, survival and quality of life and patients previously diagnosed with stage IV NSCLC within one year prior to initiating the study, (n=300).

1b. Establish a cohort of newly diagnosed stage IV non-small cell lung cancer patients (NSCLC), documenting usual care (UC) practices, survival and quality of life and patients previously diagnosed with stage IV NSCLC within one year prior to initiating the study, (n=800). This cohort will be limited to subjects directly recruited from Ohio State University for the duration of the study.

2. Following the 3 month observation period, conduct a two-phase, cluster-randomized 21 month clinical trial in stage IV NSCLC patients (n=2100).

Phase 1: Over 9 months, sites will be randomized to offer patients either UC (70% of sites) or free advanced genomic and immunotherapy testing (AGIT) (next generation sequencing tumor or blood circulating tumor DNA and PD-L1 testing immunohistochemistry staining, 30% of sites), followed by medical record review and recontacting of patients, (n=900).

Phase 2: Over 12 months, sites will be randomized to offer patients AGIT or AGIT with decision support (DS) through a genomics board, followed by medical record review and recontacting of patients, (n=1200).

3. Following the Aim 1 three month observation period, for subjects enrolled in Aim 2 (both phases) who smoke or have recently quit smoking (n=336), and their household members who smoke (n=84), to conduct a 1 year smoking cessation intervention trial where subjects are randomized by site to receive UC or National Cancer Center Network (NCCN)-driven centralized telephone counseling and decision support (CTC/DS).

4. Separately, we will identify epigenetic biomarkers as prognostic and predictive biomarkers and analyze immune profile as biomarkers for immune-related adverse events. Assays will be performed using samples and data from subjects who consent to the repository.

4a. We will identify tumor epigenetic biomarkers (DNA methylation by Illumina methylation profiling) for immunotherapy (IOT) response in stage IV NSCLC (n=50 participants each with PD-L1 expression <1% and >50%) and extend the results to the study of blood cell-free DNA (cfDNA).

4b. We will identify immune profile using blood transcriptomics as biomarkers for IOT Immune-Related Adverse Events (irAE) (n=50).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I (UC): Patients receive usual care and undergo collection of tumor tissue and blood sample for the repository. Patients who smoke or have recently quit smoking and their household members who smoke may also undergo smoking cessation via usual care or NCCN driven-CTC/DS.

ARM II (AGIT/DS): Patients undergo collection of tumor tissue for analysis using FoundationOne assay and blood sample for analysis using FoundationACT blood circulating tumor DNA assay. Patients who smoke or have recently quit smoking and their household members who smoke may also undergo smoking cessation via usual care or NCCN driven-CTC/DS.

ELIGIBILITY:
Inclusion Criteria:

* AIM 1-3
* Pathologically confirmed stage IV NSCLC (with any Eastern Cooperative Oncology Group [ECOG] performance status, and any NSCLC - adenocarcinoma, squamous cell, etc.) with available imaging OR patients who do not yet have their staging completed, but in the judgment of the physician are likely to be stage IV;

  * Patients may be enrolled if the recruiter cannot reach the patient by the first office visit, preferably prior to starting therapy and no later than one month after starting therapy; (NCCN guidelines allow for a switch to targeted therapy from chemotherapy if testing comes back positive after starting chemotherapy)
* English speaking; and
* Willing to provide access to medical records, insurance and billing data, biospecimens and respond to questionnaires, typically by phone, but possibly to include online or in-person surveys
* AIM 3 ONLY
* Patients must be current smokers who smoke at least one cigarette most days per week, or recent quitters who smoked at least one cigarette most days per week (< 3 months); and
* Household members must be current smokers, defined as smoking at least one cigarette most days per week
* Hearing and vision impairments that would prevent ability to complete consent, interviews, or sample collection

Exclusion Criteria:

* Being treated with definitive chemoradiotherapy or surgery
* Receiving treatment for advanced lung cancer for over one month before enrollment; OR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3584 (Estimated)
Dates: Start 2017-07-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Cost-Effectiveness Analysis | Up to 24 months
  Using the payer perspective, Incremental Cost-Effectiveness Ratio (ICER) will be calculated based on estimates of overall survival/health care resource costs associated with treatment and the EQ5D questionnaire.
Overall survival (Aim I observational phase) | Up to 3 years
  Descriptive statistics (summaries, distributions, 95% confidence intervals) will be reported and compared with the two arms in the randomized trial phase. Graphical displays will be used to show distributions (boxplots, density curves) and Kaplan-Meier plots to display survival curves.
Percent of patients receiving first line targeted therapy (Aim I observational phase) | Up to 3 years
  Descriptive statistics (summaries, distributions, 95% confidence intervals) will be reported and compared with the two arms in the randomized trial phase. Graphical displays will be used to show distributions (boxplots, density curves).
Percent of patients receiving genomic testing at diagnosis and type of genomic testing (Aim I observational phase) | Up to 3 years
  Descriptive statistics (summaries, distributions, 95% confidence intervals) will be reported and compared with the two arms in the randomized trial phase. Graphical displays will be used to show distributions (boxplots, density curves).
Percent of patients receiving genomic testing later in treatment (Aim I observational phase) | Up to 3 years
  Descriptive statistics (summaries, distributions, 95% confidence intervals) will be reported and compared with the two arms in the randomized trial phase. Graphical displays will be used to show distributions (boxplots, density curves).
Percent of patients receiving off label therapy (Aim I observational phase) | Up to 3 years
  Descriptive statistics (summaries, distributions, 95% confidence intervals) will be reported and compared with the two arms in the randomized trial phase. Graphical displays will be used to show distributions (boxplots, density curves).
Percent of patients referred to clinical trials (Aim I observational phase) | Up to 3 years
  Descriptive statistics (summaries, distributions, 95% confidence intervals) will be reported and compared with the two arms in the randomized trial phase. Graphical displays will be used to show distributions (boxplots, density curves) and Kaplan-Meier plots to display survival curves.
Percent of patients who enroll in therapeutic clinical trials (Aim I observational phase) | Up to 3 years
  Descriptive statistics (summaries, distributions, 95% confidence intervals) will be reported and compared with the two arms in the randomized trial phase. Graphical displays will be used to show distributions (boxplots, density curves).
Progression free survival (Aim I observational phase) | Up to 3 years
  Descriptive statistics (summaries, distributions, 95% confidence intervals) will be reported and compared with the two arms in the randomized trial phase. Graphical displays will be used to show distributions (boxplots, density curves) and Kaplan-Meier plots to display survival curves.
Quality of life assessed using European Organization for Research and Treatment-quality of life questionnaire | Up to 24 months
  For aim II, a linear mixed model will be used to model change in quality of life as subjects are transitioned from one therapy to the next, with a main effect for treatment group and random effect for hospital and patient nested within hospital. To allow for possible changes in trajectories over time (e.g., a change-point analysis) the 'segmented' package in R will be used. Trajectories for each treatment will be modeled using a segmented mixed model with random change points as implemented in R. Variables associated with missing values will be evaluated and potentially included in the mixed m
Smoking cessation (Aim III centralized telephone counseling/decision support) | Up to 6 months
  Primary analysis will focus on smoking cessation at six months follow-up using generalized linear mixed models with a random effect for practice. The odds ratio and 95% confidence interval between smoking cessation and intervention arm will be reported based on the generalized linear mixed models model. As an alternative, we will also fit competing risks regression models (e.g., using the R package 'cmprsk') with death and smoking cessation as competing events. Subdistribution function hazard ratios for smoking cessation based on the intervention will be reported.
Survival (Aim 2 advanced genomic and immunotherapy testing/decision support) | Up to 3 years
  Overall differences in survival between the advanced genomic and immunotherapy testing and usual care arms will be assessed using the log-rank test. Cox proportional hazards model will be fit with a random effect for hospital and time to obtain the hazard ratio and 95% confidence interval for the treatment effect (advanced genomic and immunotherapy testing versus usual care). Interaction between treatment and time (e.g., via a time-dependent treatment effect) will be evaluated to assess possible evolution in usual care over time. To assess clinical decision making and clinical trial referral.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Shields, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park KR, Shields PG, Myers JV, Reisinger SA, Andersen BL. Depression and Inflammation Predict Depression Trajectory of Non-Small Cell Lung Cancer Patients. Biopsychosoc Sci Med. 2025 Jul-Aug 01;87(6):397-404. doi: 10.1097/PSY.0000000000001379. Epub 2025 Jun 11. PMID 40511978
- [Derived] Valentine TR, Park KR, Presley CJ, Shields PG, Andersen BL. Lung cancer patients' illness perceptions: Prognostic for psychological and physical health trajectories. Health Psychol. 2024 Dec;43(12):913-923. doi: 10.1037/hea0001416. Epub 2024 Sep 26. PMID 39325429
- [Derived] Blevins TR, Lo SB, Coker CA, Arrato NA, Reisinger SA, Shields PG, Andersen BL. COVID-19 or Cancer Stress? Anxiety and Depressive Symptoms in Patients with Advanced Lung Cancer. Int J Behav Med. 2024 Apr;31(2):325-330. doi: 10.1007/s12529-023-10206-w. Epub 2023 Aug 18. PMID 37594667
- [Derived] Andersen BL, Myers J, Blevins T, Park KR, Smith RM, Reisinger S, Carbone DP, Presley CJ, Shields PG, Carson WE. Depression in association with neutrophil-to-lymphocyte, platelet-to-lymphocyte, and advanced lung cancer inflammation index biomarkers predicting lung cancer survival. PLoS One. 2023 Feb 24;18(2):e0282206. doi: 10.1371/journal.pone.0282206. eCollection 2023. PMID 36827396
- [Derived] Valentine TR, Presley CJ, Carbone DP, Shields PG, Andersen BL. Illness perception profiles and psychological and physical symptoms in newly diagnosed advanced non-small cell lung cancer. Health Psychol. 2022 Jun;41(6):379-388. doi: 10.1037/hea0001192. PMID 35604701
- [Derived] Arrato NA, Lo SB, Coker CA, Covarrubias JJ, Blevins TR, Reisinger SA, Presley CJ, Shields PG, Andersen BL. Cancer Treatment During COVID-19: Resilience of Individuals With Advanced Non-Small Cell Lung Cancer Versus Community Controls. J Natl Compr Canc Netw. 2022 Feb;20(2):118-125. doi: 10.6004/jnccn.2021.7076. PMID 35130505
- [Derived] Andersen BL, McElroy JP, Carbone DP, Presley CJ, Smith RM, Shields PG, Brock GN. Psychological Symptom Trajectories and Non-Small Cell Lung Cancer Survival: A Joint Model Analysis. Psychosom Med. 2022 Feb-Mar 01;84(2):215-223. doi: 10.1097/PSY.0000000000001027. PMID 34629425
- [Derived] Andersen BL, Valentine TR, Lo SB, Carbone DP, Presley CJ, Shields PG. Newly diagnosed patients with advanced non-small cell lung cancer: A clinical description of those with moderate to severe depressive symptoms. Lung Cancer. 2020 Jul;145:195-204. doi: 10.1016/j.lungcan.2019.11.015. Epub 2019 Nov 21. PMID 31806360
- See also: The Jamesline — http://cancer.osu.edu